CLINICAL TRIAL: NCT06505200
Title: An Integrative Clinicopathological Decision Support System for Kidney Transplant Rejection
Brief Title: Observational Cohort Study Renal Transplantation University Hospitals Leuven
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64006
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant Rejection; Kidney Transplantation; Kidney Transplant Failure
Keywords: Clinical Decision Support; Outcome; Risk Markers; Stratification; Histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This observational cohort study aims to compile routinely collected clinical, histological and outcome data of kidney transplant recipients, to evaluate risk factors for post-transplant injury, phenotypes of injury, and impact on outcome of such injury, in order to provide clinicians more accurate, less biased and faster tools for diagnosis, clinical management and treatment decisions with regard to kidney transplant rejection.

DETAILED DESCRIPTION:
The following data/features are collected prospectively and structured in the electronic medical records:

Demographics:

* Date of transplantation
* Date of graft failure
* Last date of follow-up
* Time after transplantation of survival (number of days);
* kidney survival;
* recipient death;
* recipient gender;
* recipient age at time of transplantation;
* recipient weight at time of transplantation;
* recipient BMI at time of transplantation;
* recipient race;
* recipient diabetes prior to transplantation;
* the Belgian Index for Multiple Deprivation (BIMD);
* combined vs single transplant (we included only single transplants);
* repeat transplant vs. first transplant;
* diagnosis of the original kidney disease (prior to transplantation);
* donor type (living vs. deceased);
* donor gender;
* donor age in years;
* donor diabetes yes vs no;
* HLA genotype of donors and recipients, number of HLA A mismatches between donor and recipient (0-2); number of HLA B mismatches between donor and recipient (0-2); number of HLA DR mismatches between donor and recipient (0-2); number of total HLA mismatches between donor and recipient (0-6); high-resolution genotyping of donors and recipients HLA genes (11 loci);
* cold ischemia time
* warm ischemia time
* operation time

Graft functional data:

* Serum creatinine values from day of transplantation onwards;
* Proteinuria values from day of transplantation onwards

Data on DSA:

DSA data collected in clinical routine, from the day of listing for transplantation onwards (clinically measured at the Histocompatibility laboratory of the Red Cross, Motstraat, Mechelen, and reported in the clinical patient records).

Biopsy data:

Both clinically indicated and protocol biopsies were performed in this cohort. On average, 3.2 biopsies per patient.

* The following data are collected from the clinical records and transferred to a pseudonymized database: Date of the kidney biopsy; Indication biopsy = at time of graft dysfunction; protocol = prespecified biopsy per protocol; pretransplant = biopsy prior to transplantation (in the donor); post-transplant = biopsy after transplantation; time point (indication vs. Protocol biopsy time points); tubulitis (0-3); interstitial inflammation (0-3); vasculitis (0-3); glomerulitis (0-3); peritubular capillaritis (0-3); thrombi (0-3); C4d deposition in peritubular capillaries (0-3); C4d deposition in glomerular capillaries (0-3); transplant glomerulopathy (0-3); interstitial fibrosis (0-3); tubular atrophy (0-3); vascular intimal thickening (0-3); mesangial matrix increase (0-3); arteriolar hyalinosis (0-3); glomerulosclerosis (%); microcirculatory inflammation (0-6) = g + ptc; diagnosis of antibody-mediated rejection yes vs no according to current international consensus, calculated from g, ptc, cg, thrombi, C4d_ptc and v; diagnosis of T-cell mediated rejection yes vs no according to current international consensus (0 = absent, 1 = borderline; 1=present); diagnosis of IFTA grade (0-3) according to current international consensus: calculated from ci and ct
* Next to pseudonymized clinical data, also histological slides are retrieved from the biobank of the Department of Pathology of the University Hospitals Leuven and whole slide images made available for image analysis.

ELIGIBILITY:
Inclusion Criteria:

* All adult kidney transplant recipients transplanted at the University Hospitals Leuven between 01/03/2004 and 01/06/2022, without restrictions with regard to age, sex, underlying kidney disease etc.

Exclusion Criteria:

* Patients with combined transplantations (e.g. heart + kidney, liver + kidney, lung + kidney)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All renal allograft recipients transplanted at the University Hospitals Leuven between 01/03/2004 and 01/06/2022 are included in this study, without restrictions with regard to age, sex, underlying kidney disease etc.
Sampling Method: Non-Probability Sample
Enrollment: 1891 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Kidney transplant failure | 2004 - 2022
  Graft failure, recipient death

SECONDARY OUTCOMES:
Kidney transplant rejection phenotypes | 2004 - 2022
Kidney transplant function | 2004 - 2022

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Naesens, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data can only be made available to other researchers with a dedicated data transfer agreement.

REFERENCES:
- [Background] Cleenders E, Coemans M, Meziyerh S, Callemeyn J, Emonds MP, Gwinner W, Kers J, Kuypers D, Scheffner I, Senev A, Van Loon E, Wellekens K, de Vries APJ, Verbeke G, Naesens M. An observational cohort study examined the change point of kidney function stabilization in the initial period after transplantation. Kidney Int. 2024 Sep;106(3):508-521. doi: 10.1016/j.kint.2024.05.030. Epub 2024 Jun 28. PMID 38945395
- [Background] Debyser T, Callemeyn J, Coemans M, Kerkhofs J, Koshy P, Kuypers D, Senev A, Tambur AR, Van Loon E, Wellekens K, Naesens M, Emonds MP. Sensitive HLA antibody testing and the risk of antibody-mediated rejection and graft failure. HLA. 2024 Jun;103(6):e15586. doi: 10.1111/tan.15586. PMID 38932739
- [Background] Yoo D, Divard G, Raynaud M, Cohen A, Mone TD, Rosenthal JT, Bentall AJ, Stegall MD, Naesens M, Zhang H, Wang C, Gueguen J, Kamar N, Bouquegneau A, Batal I, Coley SM, Gill JS, Oppenheimer F, De Sousa-Amorim E, Kuypers DRJ, Durrbach A, Seron D, Rabant M, Van Huyen JD, Campbell P, Shojai S, Mengel M, Bestard O, Basic-Jukic N, Juric I, Boor P, Cornell LD, Alexander MP, Toby Coates P, Legendre C, Reese PP, Lefaucheur C, Aubert O, Loupy A. A Machine Learning-Driven Virtual Biopsy System For Kidney Transplant Patients. Nat Commun. 2024 Jan 16;15(1):554. doi: 10.1038/s41467-023-44595-z. PMID 38228634
- [Background] Yi Z, Xi C, Menon MC, Cravedi P, Tedla F, Soto A, Sun Z, Liu K, Zhang J, Wei C, Chen M, Wang W, Veremis B, Garcia-Barros M, Kumar A, Haakinson D, Brody R, Azeloglu EU, Gallon L, O'Connell P, Naesens M, Shapiro R, Colvin RB, Ward S, Salem F, Zhang W. A large-scale retrospective study enabled deep-learning based pathological assessment of frozen procurement kidney biopsies to predict graft loss and guide organ utilization. Kidney Int. 2024 Feb;105(2):281-292. doi: 10.1016/j.kint.2023.09.031. Epub 2023 Nov 3. PMID 37923131
- [Background] Cleenders E, Koshy P, Van Loon E, Lagrou K, Beuselinck K, Andrei G, Crespo M, De Vusser K, Kuypers D, Lerut E, Mertens K, Mineeva-Sangwo O, Randhawa P, Senev A, Snoeck R, Sprangers B, Tinel C, Van Craenenbroeck A, van den Brand J, Van Ranst M, Verbeke G, Coemans M, Naesens M. An observational cohort study of histological screening for BK polyomavirus nephropathy following viral replication in plasma. Kidney Int. 2023 Nov;104(5):1018-1034. doi: 10.1016/j.kint.2023.07.025. Epub 2023 Aug 19. PMID 37598855
- [Background] Truchot A, Raynaud M, Kamar N, Naesens M, Legendre C, Delahousse M, Thaunat O, Buchler M, Crespo M, Linhares K, Orandi BJ, Akalin E, Pujol GS, Silva HT Jr, Gupta G, Segev DL, Jouven X, Bentall AJ, Stegall MD, Lefaucheur C, Aubert O, Loupy A. Machine learning does not outperform traditional statistical modelling for kidney allograft failure prediction. Kidney Int. 2023 May;103(5):936-948. doi: 10.1016/j.kint.2022.12.011. Epub 2022 Dec 23. PMID 36572246
- [Background] Vaulet T, Divard G, Thaunat O, Koshy P, Lerut E, Senev A, Aubert O, Van Loon E, Callemeyn J, Emonds MP, Van Craenenbroeck A, De Vusser K, Sprangers B, Rabeyrin M, Dubois V, Kuypers D, De Vos M, Loupy A, De Moor B, Naesens M. Data-Driven Chronic Allograft Phenotypes: A Novel and Validated Complement for Histologic Assessment of Kidney Transplant Biopsies. J Am Soc Nephrol. 2022 Nov;33(11):2026-2039. doi: 10.1681/ASN.2022030290. Epub 2022 Sep 7. PMID 36316096
- [Background] Coemans M, Verbeke G, Dohler B, Susal C, Naesens M. Bias by censoring for competing events in survival analysis. BMJ. 2022 Sep 13;378:e071349. doi: 10.1136/bmj-2022-071349. No abstract available. PMID 36100269
- [Background] Senev A, Van Loon E, Lerut E, Coemans M, Callemeyn J, Daniels L, Kerkhofs J, Koshy P, Kuypers D, Lamarthee B, Sprangers B, Tinel C, Van Craenenbroeck AH, Van Sandt V, Emonds MP, Naesens M. Association of Predicted HLA T-Cell Epitope Targets and T-Cell-Mediated Rejection After Kidney Transplantation. Am J Kidney Dis. 2022 Dec;80(6):718-729.e1. doi: 10.1053/j.ajkd.2022.04.009. Epub 2022 Jun 9. PMID 35690154
- [Background] Senev A, Lerut E, Coemans M, Callemeyn J, Copley HC, Claas F, Koshy P, Kosmoliaptsis V, Kuypers D, Sprangers B, Van Craenenbroeck A, Van Loon E, Van Sandt V, Emonds MP, Naesens M. Association of HLA Mismatches and Histology Suggestive of Antibody-Mediated Injury in the Absence of Donor-Specific Anti-HLA Antibodies. Clin J Am Soc Nephrol. 2022 Aug;17(8):1204-1215. doi: 10.2215/CJN.00570122. Epub 2022 Jun 1. PMID 35649719
- [Background] Van Loon E, Zhang W, Coemans M, De Vos M, Emonds MP, Scheffner I, Gwinner W, Kuypers D, Senev A, Tinel C, Van Craenenbroeck AH, De Moor B, Naesens M. Forecasting of Patient-Specific Kidney Transplant Function With a Sequence-to-Sequence Deep Learning Model. JAMA Netw Open. 2021 Dec 1;4(12):e2141617. doi: 10.1001/jamanetworkopen.2021.41617. PMID 34967877
- [Background] Kers J, Bulow RD, Klinkhammer BM, Breimer GE, Fontana F, Abiola AA, Hofstraat R, Corthals GL, Peters-Sengers H, Djudjaj S, von Stillfried S, Holscher DL, Pieters TT, van Zuilen AD, Bemelman FJ, Nurmohamed AS, Naesens M, Roelofs JJTH, Florquin S, Floege J, Nguyen TQ, Kather JN, Boor P. Deep learning-based classification of kidney transplant pathology: a retrospective, multicentre, proof-of-concept study. Lancet Digit Health. 2022 Jan;4(1):e18-e26. doi: 10.1016/S2589-7500(21)00211-9. Epub 2021 Nov 15. PMID 34794930
- [Background] Callemeyn J, Senev A, Coemans M, Lerut E, Sprangers B, Kuypers D, Koenig A, Thaunat O, Emonds MP, Naesens M. Missing Self-Induced Microvascular Rejection of Kidney Allografts: A Population-Based Study. J Am Soc Nephrol. 2021 Aug;32(8):2070-2082. doi: 10.1681/ASN.2020111558. Epub 2021 Jul 22. PMID 34301794
- [Background] Coemans M, Senev A, Van Loon E, Lerut E, Sprangers B, Kuypers D, Emonds MP, Verbeke G, Naesens M. The evolution of histological changes suggestive of antibody-mediated injury, in the presence and absence of donor-specific anti-HLA antibodies. Transpl Int. 2021 Oct;34(10):1824-1836. doi: 10.1111/tri.13964. Epub 2021 Sep 12. PMID 34197662
- [Background] Senev A, Emonds MP, Naesens M. Second field high-resolution HLA typing for immunologic risk stratification in kidney transplantation. Am J Transplant. 2021 Oct;21(10):3502-3503. doi: 10.1111/ajt.16606. Epub 2021 Apr 30. No abstract available. PMID 33866671
- [Background] Vaulet T, Divard G, Thaunat O, Lerut E, Senev A, Aubert O, Van Loon E, Callemeyn J, Emonds MP, Van Craenenbroeck A, De Vusser K, Sprangers B, Rabeyrin M, Dubois V, Kuypers D, De Vos M, Loupy A, De Moor B, Naesens M. Data-driven Derivation and Validation of Novel Phenotypes for Acute Kidney Transplant Rejection using Semi-supervised Clustering. J Am Soc Nephrol. 2021 May 3;32(5):1084-1096. doi: 10.1681/ASN.2020101418. Epub 2021 Mar 9. PMID 33687976
- [Background] Senev A, Van Loon E, Lerut E, Callemeyn J, Coemans M, Van Sandt V, Kuypers D, Emonds MP, Naesens M. Risk factors, histopathological features, and graft outcome of transplant glomerulopathy in the absence of donor-specific HLA antibodies. Kidney Int. 2021 Aug;100(2):401-414. doi: 10.1016/j.kint.2021.01.029. Epub 2021 Mar 3. PMID 33675843
- [Background] Reese PP, Aubert O, Naesens M, Huang E, Potluri V, Kuypers D, Bouquegneau A, Divard G, Raynaud M, Bouatou Y, Vo A, Glotz D, Legendre C, Lefaucheur C, Jordan S, Empana JP, Jouven X, Loupy A. Assessment of the Utility of Kidney Histology as a Basis for Discarding Organs in the United States: A Comparison of International Transplant Practices and Outcomes. J Am Soc Nephrol. 2021 Feb;32(2):397-409. doi: 10.1681/ASN.2020040464. Epub 2020 Dec 15. PMID 33323474
- [Background] Koenig A, Mezaache S, Callemeyn J, Barba T, Mathias V, Sicard A, Charreau B, Rabeyrin M, Dijoud F, Picard C, Meas-Yedid V, Olivo-Marin JC, Morelon E, Naesens M, Dubois V, Thaunat O. Missing Self-Induced Activation of NK Cells Combines with Non-Complement-Fixing Donor-Specific Antibodies to Accelerate Kidney Transplant Loss in Chronic Antibody-Mediated Rejection. J Am Soc Nephrol. 2021 Feb;32(2):479-494. doi: 10.1681/ASN.2020040433. Epub 2020 Nov 25. PMID 33239394
- [Background] Raynaud M, Aubert O, Reese PP, Bouatou Y, Naesens M, Kamar N, Bailly E, Giral M, Ladriere M, Le Quintrec M, Delahousse M, Juric I, Basic-Jukic N, Gupta G, Akalin E, Yoo D, Chin CS, Proust-Lima C, Bohmig G, Oberbauer R, Stegall MD, Bentall AJ, Jordan SC, Huang E, Glotz D, Legendre C, Montgomery RA, Segev DL, Empana JP, Grams ME, Coresh J, Jouven X, Lefaucheur C, Loupy A. Trajectories of glomerular filtration rate and progression to end stage kidney disease after kidney transplantation. Kidney Int. 2021 Jan;99(1):186-197. doi: 10.1016/j.kint.2020.07.025. Epub 2020 Aug 8. PMID 32781106
- [Background] Van Loon E, Lerut E, Senev A, Coemans M, Pirenne J, Monbaliu D, Jochmans I, Sainz Barriga M, De Vusser K, Van Craenenbroeck AH, Sprangers B, Emonds MP, Kuypers D, Naesens M. The Histological Picture of Indication Biopsies in the First 2 Weeks after Kidney Transplantation. Clin J Am Soc Nephrol. 2020 Oct 7;15(10):1484-1493. doi: 10.2215/CJN.04230320. Epub 2020 Aug 10. PMID 32778537
- [Background] Senev A, Coemans M, Lerut E, Van Sandt V, Kerkhofs J, Daniels L, Driessche MV, Compernolle V, Sprangers B, Van Loon E, Callemeyn J, Claas F, Tambur AR, Verbeke G, Kuypers D, Emonds MP, Naesens M. Eplet Mismatch Load and De Novo Occurrence of Donor-Specific Anti-HLA Antibodies, Rejection, and Graft Failure after Kidney Transplantation: An Observational Cohort Study. J Am Soc Nephrol. 2020 Sep;31(9):2193-2204. doi: 10.1681/ASN.2020010019. Epub 2020 Aug 6. PMID 32764139
- [Background] Senev A, Emonds MP, Van Sandt V, Lerut E, Coemans M, Sprangers B, Kuypers D, Naesens M. Clinical importance of extended second field high-resolution HLA genotyping for kidney transplantation. Am J Transplant. 2020 Dec;20(12):3367-3378. doi: 10.1111/ajt.15938. Epub 2020 May 15. PMID 32337773
- [Background] Van Loon E, Senev A, Lerut E, Coemans M, Callemeyn J, Van Keer JM, Daniels L, Kuypers D, Sprangers B, Emonds MP, Naesens M. Assessing the Complex Causes of Kidney Allograft Loss. Transplantation. 2020 Dec;104(12):2557-2566. doi: 10.1097/TP.0000000000003192. PMID 32091487